CLINICAL TRIAL: NCT04326010
Title: Prospective Clinical Follow-up of the Echo Bi-Metric Microplasty Stem for Total Hip Arthroplasty
Status: Terminated | Type: Observational
Why Stopped: Data collected up to this point has provided sufficient follow-up and will allow for a reasonable estimate of the five-year survivorship rate for the Echo Bi-Metric Microplasty stem in primary total hip arthroplasty.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: H.CR.I.AM.16.6
Record Dates: First submitted 2020-01-24; First posted 2020-03-30 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Surgery — THA surgery

SUMMARY:
The primary objective of this study is to characterize survivorship of the Echo Bi-Metric Microplasty stem in unilateral or bilateral primary total hip arthroplasty at 5 years postoperative.

DETAILED DESCRIPTION:
Primary objective

The primary objective of this study is to characterize survivorship of the Echo Bi-Metric Microplasty stem in unilateral or bilateral primary total hip arthroplasty at 5 years postoperative.

Secondary Objectives

Safety will be evaluated by monitoring the frequency and incidence of adverse events over time to 10 years postoperative.

Clinical, functional, radiographic, and quality of life outcomes will be assessed over time to 7 years postoperative. Clinical Outcomes will be measured using the Harris Hip Score and Physical Exam form. Radiographs will be reviewed to assess alignment, radiolucencies and other radiographic parameters. Health status and functional ability will be measured using the EQ-5D-3L and the UCLA Activity score.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible for this trial if they satisfy all of the following criteria:

  * Patient is 18 to 65 years of age, inclusive
  * Patient is skeletally mature
  * Patient qualifies for primary unilateral or bilateral total hip arthroplasty based on physical exam and medical history including at least one of the following:
  * Osteoarthritis
  * Avascular necrosis
  * Rheumatoid arthritis
  * Correction of functional deformity
  * Treatment of non-union, femoral neck fracture, and trochanteric fractures of the proximal femur with head involvement, unmanageable by other techniques
  * Patient has no history of previous total hip arthroplasty or arthrodesis of the affected hip joint(s)
  * Patient is willing and able to complete scheduled follow-up evaluations as described in the Informed Consent
  * Patient, or the patient's legally authorized representative, has participated in the Informed Consent process and is willing and able to sign an IRB- approved informed consent

Exclusion Criteria:

* Subjects will be excluded from this trial if they satisfy any of the following criteria as determined by the research staff or in the judgment of the treating physician:

  * Patient has a total prosthetic hip replacement device (including surface replacement arthroplasty, endoprosthesis, etc.) in the affected hip joint(s)
  * Patient is septic or has an active infection
  * Patient is uncooperative patient or is incapable of following directions
  * Patient is diagnosed with osteoporosis
  * Patient is diagnosed with a metabolic disorder which may impair bone formation
  * Patient is diagnosed with osteomalacia
  * Patient has distant foci of infections which may spread to the implant site

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will comprise a cohort of a minimum of 200, and no more than 225, hips enrolled across up to 10 centers from subjects who require primary total hip arthroplasty. Subjects must be willing and able to attend required follow-up appointments. Candidates who express interest in study participation will undergo an informed consent procedure, be required to sign an IRB-approved informed consent with required HIPAA authorization1, and eligibility will be determined based upon the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-12-04 (Actual)

PRIMARY OUTCOMES:
Implant Survival | 5 years postoperatively / Life of Study
  The primary objective of this study is to characterize survivorship of the Echo Bi-Metric Microplasty stem in unilateral or bilateral primary total hip arthroplasty at 5 years postoperative.

SECONDARY OUTCOMES:
Clinical Outcomes | 7 Years Post-Operative.
  Clinical Outcomes will be measured using the Harris Hip Score and Physical Exam form.
Functional Outcomes | 7 Years Post-Operative
  Functional ability will be measured using the EQ-5D-3L.
Radiographic Outcomes | 7 Years Post-Operative
  Standard AP and lateral Hip radiographics of the implanted hip device will be assess the positioning of the device as well as lucencies and other potential anomalies
Quality of Life Outcomes | 7 Years Post-Operative
  Will be measured by UCLA Activity Score
Safety Outcomes | 10 Years Post-Operative
  Will be evaluated by monitoring the frequency and incidence of adverse events over time of the study

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, BS, Study Director — Zimmer Biomet
Locations (6):
- United States (6):
  - OrthoSports Associates, Birmingham, Alabama
  - University of CA - San Diego, San Diego, California
  - Southern Joint Replacement Institute, Nashville, Tennessee
  - Growth Ortho, Austin, Texas
  - Tidewater Orthpaedics, Hampton, Virginia
  - Jordan-young Institute, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: Undecided